CLINICAL TRIAL: NCT04544488
Title: Descriptive Evaluation of Expulsive Efforts During Pregnancy in Term Nulliparous Women by Measurement of Intra Bladder Pressure: Pilot Observational Study.
Acronym: ACCOUPIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ACCOUPIV
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Perineal Tear

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Recording of expulsive efforts by connection of a pressure sensor to the women's bladder probe — Using a pressure probe connected to a Foley Catheter, intra bladder pressure wille be registered during the whole duration of expulsive phase.
  The device will be inserted into women's bladder using usual guidelines for insertion of Foley catheter

SUMMARY:
Severe complications of childbirth are common. Many factors have been studied to assess their imputability in the occurrence of perineal tears. While women subjectively have different push profiles in terms of intensity, frequency and duration of each push effort, no study has evaluated this variability in a relevant, simple and reproducible way. Through this work, it is expected to establish a qualitative evaluation of the expulsive efforts during childbirth in term nulliparous women by measuring the intra bladder pressure which testifies of the pressure exerted on the perineal tissues due to maternal pushing efforts

DETAILED DESCRIPTION:
Scientific context:

It is clearly observed in clinical practice that there seems to be significant variability in the characteristics of the expulsive phase from one woman to another without this being clearly described to date. During the same expulsive phase, the number, intensity and duration of each push can be very different from one woman to another.

Considering that during expulsive efforts, the fetal head exerts pressure on the perineal tissues , the repetition of these compressions, moreover if they are prolonged or brought closer together could generate muscular lesions by hyper extension of the fibers, by microtrauma or by tissue hypoxia. These variations in the characteristics of expulsive efforts could thus modify the perineal risk for women.

More than the expulsive efforts evaluated by the recording of intra uterine pressures which has already been described, it is the evaluation of the mechanical stresses transmitted to the perineum secondary to the pushing efforts that we would like to record by the installation of a sensor pressure connected to the woman's bladder catheter.

Investigations During the second phase of labor, at 8 cm dilation, after information and obtaining free and informed consent, women will be included by one of the MD investigators.

3 visits are planned in the protocol: The first visit will be at childbirth Evaluation of the mechanical stresses transmitted to the perineum secondary to the pushing efforts by the installation of a sensor pressure connected to the woman's bladder catheter

Follow up A prospective study including nulliparous term pregnant women with 2 other visits planned at 3 months (12 to 16 weeks) and 6 months (26 to 30 weeks) after delivery, to assess secondary perineal complications

ELIGIBILITY:
* Inclusion criteria :

  * Pregnant women aged of 18 years or more
  * 37 weeks or more of pregnancy
  * Without any previous delivery (vaginal or cesarean delivery)
  * With a cephalic presentation fetus
  * With epidural analgesia at 8 cm cervical dilatation (inclusion)
* - Exclusion criteria:

  * Pathological pregnancy (intrauterine growth restriction, pre-eclampsia etc.)
  * Untreated psychiatric disorders
  * Women under judicial protection
  * Women without health insurance

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
characteristics of the pushing efforts assessed by measuring intra bladder pressur | Day of inclusion
  At inclusion it will be collect the characteristics of the pushing efforts: the intensity, the duration (total and of each effort) and the frequency of the expulsive efforts, which will be described in terms of mean and standard deviation.

SECONDARY OUTCOMES:
Perineal tear | Day of inclusion, immediately after delivery
  According the RCOG Classification
Clinical pelvic organ mobility | 12 to 16 weeks after inclusion then 26 to 30 weeks after inclusion
  POP-Q clinical examination
Ultrasound pelvic organ mobility | 12 to 16 weeks after inclusion then 26 to 30 weeks after inclusion
  Transperineal pelvic floor ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided